CLINICAL TRIAL: NCT06391359
Title: Preventing Recurrent 'Idiopathic' Acute Pancreatitis Through Laparoscopic Cholecystectomy (PICUS-2): a Multicenter Randomized Trial
Brief Title: Preventing Recurrent 'Idiopathic' Acute Pancreatitis Through Laparoscopic Cholecystectomy (PICUS-2)
Acronym: PICUS-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.G. Besselink (Other)
Responsible Party: Sponsor-Investigator, M.G. Besselink, Professor, MD PhD, Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL82531.018.23
Record Dates: First submitted 2024-01-30; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Acute Pancreatitis
MeSH Terms: interventions — Cholecystectomy, Laparoscopic; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic cholecystectomy (Experimental)
  Interventions: Procedure: Laparoscopic cholecystectomy
- Watchful waiting (Active Comparator)
  Interventions: Other: Watchful waiting

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy
  Arms: Laparoscopic cholecystectomy
Other: Watchful waiting — Watchful waiting
  Arms: Watchful waiting

SUMMARY:
Rationale: Annually, acute pancreatitis is diagnosed in 6,500 patients in the Netherlands. In up to 25% of patients no definitive cause can be determined after routine work-up including endoscopic ultrasound and this is deemed to be idiopathic acute pancreatitis (IAP). IAP is known for its high recurrence rate. It is hypothesized that microlithiasis, a type of biliary pancreatitis, is the most common cause of IAP. Laparoscopic cholecystectomy (LC) is highly effective in preventing recurrence of biliary pancreatitis. Currently no randomized trial has compared LC with conservative treatment in patients with IAP after adequate work-up including endoscopic ultrasound.

Objective: To assess the effectiveness of LC as compared to conservative treatment in patients after a first episode of 'EUS-negative' IAP.

Study design: Multicenter randomized controlled trial. Patients will be followed for one year after randomization.

Study population: Adults with a first episode of 'EUS-negative' IAP.

Intervention (if applicable): Laparoscopic cholecystectomy versus conservative treatment.

Main study parameters/endpoints: The primary endpoint is pancreatitis recurrence. Secondary endpoints include occurrence of biliary events, complications of LC, number and severity of recurrent episodes of pancreatitis, quality of life (QALY), costs (hospital and societal) and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Eligible for early (laparoscopic)* cholecystectomy
* Full required diagnostic work-up of patient has been performed, including EUS
* First episode of 'EUS-negative' IAP
* Informed consent for participation was obtained *if required open cholecystectomy is allowed

Exclusion Criteria:

* Recurrent acute pancreatitis
* Diagnosis of chronic pancreatitis
* Diagnosis of necrotizing pancreatitis
* Current pancreatic malignancy
* Prior cholecystectomy
* Documented etiology of acute pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2023-07-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Acute pancreatitis recurrence | Within 1 year after date of inclusion
  Acute pancreatitis recurrence, irrespective of etiology

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location University of Amsterdam, Amsterdam, North Holland, Netherlands